CLINICAL TRIAL: NCT02724644
Title: EN3835 for the Treatment of Edematous Fibrosclerotic Panniculopathy (Commonly Known as Cellulite)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EN3835-201
Record Dates: First submitted 2016-03-10; First posted 2016-03-31 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Edematous Fibrosclerotic Panniculopathy; Cellulite
MeSH Terms: conditions — Cellulite | interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EN3835 Active (Experimental): EN3835 0.84 mg (Collagenase Clostridium Histolyticum). Each subject can receive up to three treatment sessions. Each treatment session will be separated by approximately 21 days.
  Interventions: Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM
- EN3835 Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo Comparator

INTERVENTIONS:
Biological: COLLAGENASE CLOSTRIDIUM HISTOLYTICUM — Injectable intervention
  Other Names: Xiaflex
  Arms: EN3835 Active
Biological: Placebo Comparator
  Arms: EN3835 Placebo

SUMMARY:
The study will evaluate the safety, effectiveness, and immunogenicity of EN3835 in the treatment of adult women with Edematous Fibrosclerotic Panniculopathy (Commonly known as Cellulite).

ELIGIBILITY:
Inclusion Criteria:

* Be a female ≥18 years of age
* At Screening visit, have at least 1 quadrant with:

  * a score of 3 or 4 (moderate or severe) as reported by the subject (PR- PCSS), and
  * a score of 3 or 4 (moderate or severe) as reported by the Investigator (CR-PCSS), and
  * a Hexsel CSS score no greater than 13
* At Day 1 visit, have an assigned quadrant with:

  * a score of 3 or 4 (moderate or severe) as reported by the subject (PR-PCSS), and
  * a score of 3 or 4 (moderate or severe) as reported by the Investigator (CR-PCSS), and
  * a Hexsel CSS score no greater than 13
* Be willing to apply sunscreen to the selected treatment quadrant before each exposure to the sun while participating in the study (ie, screening through end of study).
* Be judged to be in good health, based upon the results of a medical history, physical examination, and laboratory profile at screening
* Have a negative urine pregnancy test at screening and be using an effective contraception method (eg, abstinence, intrauterine device [IUD], hormonal [estrogen/progestin] contraceptives, or double barrier method) for at least 1 menstrual cycle prior to study enrollment and for the duration of the study; or be menopausal defined as 12 months of amenorrhea in the absence of other biological or physiological causes, as determined by the investigator; or post-menopausal for at least 1 year; or be surgically sterile.
* Be willing and able to cooperate with the requirements of the study
* Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee/Human Research Ethics Committee (IRB/IEC/HREC).
* Be able to read, complete and understand the Patient Reported Outcomes rating instruments in English

Exclusion Criteria:

* Has any of the following conditions:

  * Thyroid disease, unless controlled with medication for ≥6 months
  * Uncontrolled diabetes mellitus, as determined by the Investigator
  * Uncontrolled hypertension, as determined by the Investigator
  * Vascular disorder (eg, phlebitis or varicose veins) in area to be treated
  * Cushing's disease and/or use of systemic corticosteroids at a total daily dose greater than 5 mg prednisone (or equivalent)
  * History of lower extremity thrombosis or post-thrombosis syndrome
  * Documented autoimmune disorder such as lupus erythematosus, rheumatoid arthritis
  * Inflammation or active infection in area to be treated
  * Active cutaneous alteration in area to be treated including rash, eczema, psoriasis or skin cancer
  * History of keloidal scarring or abnormal wound healing
  * Coagulation disorder
  * Taking a medication for chronic anticoagulation (except for ≤150 mg aspirin daily)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Clinical Testing of Beverly Hills, Beverly Hills, California
  - Dermatology Specialists, Inc, Murrieta, California
  - Dermatology Specialists, Inc, Oceanside, California
  - Dermatology Cosmetic Laser Medical Associates of LaJolla, Inc, San Diego, California
  - Olympian Clinical Research, Clearwater, Florida
  - Skin Research Institute LLC, Coral Gables, Florida
  - Research Institute of the Southeast, West Palm Beach, Florida
  - Mercy Health Research, Washington, Missouri
  - Bass Plastic Surgery, PLLC, New York, New York
  - Sadick Research Group, New York, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Charlottesville Medical Research Center LLC, Charlottesville, Virginia
  - The Education & Research Foundation, Lynchburg, Virginia
  - Premier Clinical Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- EN3835 0.84 mg: Three (3) treatment sessions of 0.84 mg of collagenase clostridium histolyticum separated by approximately 21 days.
  Injectable intervention
- Placebo: Three (3) treatment sessions of placebo separated by approximately 21 days. Injectable intervention
Period: Overall Study
Arm/Group | EN3835 0.84 mg | Placebo
Started | 189 | 186
Completed | 168 | 182
Not Completed | 21 | 4
Not completed — Adverse Event | 7 | 1
Not completed — Lost to Follow-up | 6 | 2
Not completed — Withdrawal by Subject | 7 | 1
Not completed — Administrative | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis based on intent-to-treat (ITT) population; all randomized subjects who received at least 1 injection of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | EN3835 0.84 mg | Placebo | Total
Number analyzed (Participants) | 189 | 186 | 375
Age, Continuous [Mean (Standard Deviation); unit: Participants] | 47.2 (11.21) | 45.8 (11.02) | 46.5 (11.13)
Age, Customized [Count of Participants; unit: Participants]
  18-<25 years | 8 | 9 | 17
  25-34 years | 18 | 21 | 39
  35-44 years | 46 | 47 | 93
  >=45 years | 117 | 109 | 226
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189 | 186 | 375
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 41 | 78
  Not Hispanic or Latino | 152 | 145 | 297
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 15 | 26 | 41
  White | 167 | 157 | 324
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 189 | 186 | 375

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Composite Responders of at Least 2-Level Improvement of Severity
Description: Percentage of composite responders defined as subjects with an improvement from baseline of at least 2-levels of severity on each, the Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS), at Day 71 in the ITT population. The CR-PCSS is a photonumeric scale that was used by the Investigator to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). The PR-PCSS is a photonumeric scale that was used by the subjects to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). A 2-level improvement on each scale for example would represent a change from a 4 (severe) to a 2 (mild). In order to be considered a responder a subject needs to have at least a 2-level improvement on both scales.
Time Frame: Baseline, Day 71
Population: Analysis is based on ITT population; all randomized subjects who received at least 1 injection of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 189 | 186
Participants | 20 | 3

2. Secondary Outcome: Percentage of Composite Responders of at Least 1-Level Improvement of Severity
Description: Percentage of composite responders defined as subjects with improvement from baseline of at least 1-level of severity on each, the Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS), at Day 71 in the ITT population. The CR-PCSS is a photonumeric scale that was used by the Investigator to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). The PR-PCSS is a photonumeric scale that was used by the subjects to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). A 1-level improvement on each scale for example would represent a change from a 4 (severe) to a 3 (moderate). In order to be considered a responder a subject needs to have at least a 1-level improvement on both scales.
Time Frame: Baseline, Day 71
Population: Analysis is based on ITT population; all randomized subjects who received at least 1 injection of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 189 | 186
Participants | 79 | 33

3. Secondary Outcome: CR-PCSS Responder Analysis: 2-Levels of Severity
Description: Percentage of subjects with improvement from baseline of at least 2-levels of severity on the Investigator-rated Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) at Day 71.The CR-PCSS is a photonumeric scale that was used by the Investigator to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). A 2-level improvement would be for example a change from 4 (severe) to 2 (mild).
Time Frame: Baseline, Day 71
Population: Analysis is based on modified intent-to-treat (mITT) population; all randomized subjects who received at least 1 injection of study medication and had at least 1 post-injection evaluation of both CR-PCSS by investigator and PR PCSS
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
Participants | 32 | 9

4. Secondary Outcome: CR-PCSS Responder Analysis: 1-Level of Severity
Description: Percentage of subjects with improvement from baseline of at least 1-level of severity on the Investigator-rated Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) at Day 71.The CR-PCSS is a photonumeric scale that was used by the investigator to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). A 1-level improvement would be for example a change from 4 (severe) to 3 (moderate).
Time Frame: Baseline, Day 71
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
Participants | 96 | 53

5. Secondary Outcome: CR-PCSS Change From Baseline
Description: The CR-PCSS is a photonumeric scale that was used by the investigator to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). Change is Day 71 study visit rating minus baseline visit; negative values indicate a lessening in cellulite severity.
Time Frame: Baseline, Day 71
Population: Analysis is based on mITT population; all randomized subjects who received at least 1 injection of study medication and had at least 1 post-injection evaluation of both CR-PCSS by investigator and PR PCSS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
units on a scale | -0.7 (0.83) | -0.3 (0.62)

6. Secondary Outcome: PR-PCSS Responder Analysis: 2-Levels of Severity
Description: Percentage of subjects with improvement from baseline of at least 2-levels of severity on the subject-rated Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) at Day 71.The PR-PCSS is a photonumeric scale that was used by the subject to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). A 2-level improvement would be for example a change from 4 (severe) to 2 (mild).
Time Frame: Baseline, Day 71
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
Participants | 51 | 24

7. Secondary Outcome: PR-PCSS Responder Analysis: 1-Level of Severity
Description: Percentage of subjects with improvement from baseline of at least 1-level of severity on the subject-rated Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) at Day 71.The PR-PCSS is a photonumeric scale that was used by the subject to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). A 1-level improvement would be for example a change from 4 (severe) to 3 (moderate).
Time Frame: Baseline, Day 71
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
Participants | 128 | 95

8. Secondary Outcome: PR-PCSS Change From Baseline
Description: The PR-PCSS is a photonumeric scale that was used by the subjects to evaluate cellulite ranging from 0 (none), 1 (almost none), 2 (mild), 3 (moderate), to 4 (severe). Change is Day 71 study visit rating minus baseline visit; negative values indicate a lessening in cellulite severity.
Time Frame: Baseline, Day 71
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
units on a scale | -1.0 (0.89) | -0.7 (0.79)

9. Secondary Outcome: Investigator Assessment of Improvement Based on the Investigator Global Aesthetic Improvement Scale (I-GAIS)
Description: On Day 71, the Investigator determined the degree of improvement from baseline in the treated area using the 7-point I-GAIS. Ratings could be improved (+1), much improved (+2), or very much improved (+3), or no change (0), or worse (-1), much worse (-2) or very much worse (-3).
Time Frame: Day 71
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
Participants
  Very Much Improved (3) | 6 | 2
  Much improved (2) | 40 | 15
  Improved (1) | 64 | 43
  No Change( 0) | 57 | 119
  Worse (-1) | 6 | 4
  Much worse (-2) | 2 | 0
  Very Much Worse (-3) | 0 | 0
  Not done | 2 | 1

10. Secondary Outcome: Subject Assessment of Improvement Based on the Subject Global Aesthetic Improvement Scale (S-GAIS)
Description: At Day 71, subjects were asked to rate their opinion of the overall improvement of their treated area using the 7-point S-GAIS. Ratings could be improved (+1), much improved (+2), or very much improved (+3), or no change (0), or worse (-1), much worse (-2) or very much worse (-3)
Time Frame: Day 71
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
Participants
  Very Much Improved (3) | 21 | 11
  Much Improved (2) | 43 | 17
  Improved (1) | 64 | 52
  No change (0) | 38 | 97
  Worse (-1) | 6 | 5
  Much Worse (-2) | 3 | 0
  Very Much Worse (-3) | 0 | 0
  Not done | 2 | 2

11. Secondary Outcome: Subject Satisfaction Assessment Based on the the Subject Satisfaction Scale
Description: At Day 71, subjects were asked to rate their satisfaction with cellulite treatment using the 5-point subject satisfaction scale. Ratings could be satisfied (+1), very satisfied (+2), neither satisfied nor dissatisfied (0), or dissatisfied (-1), very dissatisfied (-2).
Time Frame: Day 71
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
Participants
  Very Satisfied (2) | 41 | 25
  Satisfied (1) | 69 | 40
  Neither Satisfied nor Dissatisfied (0) | 45 | 82
  Dissatisfied (-1) | 11 | 18
  Very Dissatisfied (-2) | 9 | 16
  Not done | 2 | 3

12. Secondary Outcome: Change in the Hexsel Cellulite Severity Scale (CSS) Total Score
Description: Investigator used the Hexsel CSS to assess the severity of cellulite. The total score could range from 0 (no cellulite) to 15 (extremely severe cellulite). Negative change in Hexsel CSS total score indicates an improvement in cellulite severity
Time Frame: Baseline, Day 71
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 177 | 184
units on a scale | -1.7 (2.20) | -0.9 (2.00)

ADVERSE EVENTS:
Time Frame: Baseline, Day 71
Description: Serious Adverse Events by Frequency (Safety Population)
Arm/Group | EN3835 0.84 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/189 | 0/186
Other Adverse Events (participants affected / at risk) | 148/189 | 30/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EN3835 0.84 mg (N=189) | Placebo (N=186)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Serious Adverse Events by Frequency (Safety Population)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EN3835 0.84 mg (N=189) | Placebo (N=186)
Injection site bruising (General disorders) | 142 (314) | 25 (33) — Administration site conditions
Injection site pain (General disorders) | 112 (228) | 10 (11) — Administration site conditions
Injection site nodule (General disorders) | 27 (33) | 0 (0) — Administration site conditions
Injection site pruritus (General disorders) | 21 (29) | 1 (1) — Administration site conditions
Injection site induration (General disorders) | 11 (17) | 0 (0) — Administration site conditions
Injection site swelling (General disorders) | 14 (17) | 1 (2) — Administration site conditions
Injection site mass (General disorders) | 10 (12) | 1 (1) — Administration site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other